CLINICAL TRIAL: NCT01224769
Title: A Retrospective Multicenter Trial on Efficacy and Toxicity of Bendamustine Alone or Associated With Rituximab, as Salvage Therapy in Patients With Chronic Lymphoproliferative Disorders
Brief Title: Bendamustine and Rituximab As Salvage Therapy In Patients With Chronic Lymphoproliferative Disorders
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Studio Linfomi (Other)
Other Study IDs: RETRO-BENDA
Record Dates: First submitted 2010-10-07; First posted 2010-10-20 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2010-10

CONDITIONS: Relapsed or Refractory Chronic Lymphoproliferative Disorders
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- bendamustine +/- rituximab
  Interventions: Drug: bendamustine +/- rituximab

INTERVENTIONS:
Drug: bendamustine +/- rituximab

SUMMARY:
This retrospective study collects and evaluates the clinical experience reached in Italy on the use of bendamustine alone or combined with rituximab as treatment of patients with relapsed or refractory chronic lymphoproliferative disorders.

ELIGIBILITY:
Inclusion Criteria:

* patients with relapsed or refractory chronic lymphoproliferative disorders
* salvage treatment with bendamustine +/- rituximab
* age ≥ 18 years

Exclusion Criteria:

* previous treatment with bendamustine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with relapsed or refractory chronic lymphoproliferative disorders treated with bendamustine +/- rituximab
Sampling Method: Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2005-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
overall response rate | within 1 month after end of treatment

SECONDARY OUTCOMES:
grade III and IV (NCI Common Toxicity Criteria) adverse events | within 1 month after end of treatment
prognostic factors | within 1 month after end of treatment
progression free survival | within 1 month after end of treatment
overall survival | within 1 month after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Iannitto, MD, Study Chair — Gruppo Italiano Studio Linfomi; Fortunato Morabito, MD, Study Director — Gruppo Italiano Studio Linfomi; Stefano Luminari, MD, Principal Investigator — Gruppo Italiano Studio Linfomi
Locations (1):
- Gruppo Italiano Studio Linfomi, Modena, Italy